CLINICAL TRIAL: NCT00174382
Title: An Open-Label Trial Of Donepezil in Vascular and Mixed Dementia
Brief Title: Vaspect Study - An Open-Label Trial Of Donepezil in Vascular and Mixed Dementia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See Detailed Description
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trials Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A2501026
Record Dates: First submitted 2005-09-08; First posted 2005-09-15 (Estimated); Results first posted 2009-06-12 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Dementia, Vascular; Dementia, Mixed
MeSH Terms: conditions — Dementia, Vascular; Mixed Dementias | interventions — Donepezil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Donepezil

INTERVENTIONS:
Drug: Donepezil — donepezil 5mg/day for 6 weeks and then 5 to 10mg/day for 18 weeks

SUMMARY:
To document effectiveness, safety, and tolerability of donepezil in patients with mixed AD/VaD, and to further document the effectiveness, safety, and tolerability of donepezil in patients with VaD. The effects of donepezil on executive functioning, behavior, general cognition, ADLs and global functioning will be assessed.

DETAILED DESCRIPTION:
The trial was terminated on October 15, 2007 due to difficulties in recruiting the subjects. There were no safety or efficacy concerns regarding the study medication in the decision to terminate the trial.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet DSM-IV-TR criteria for the clinical diagnosis of Vascular Dementia or the clinical diagnosis of dementia due to multiple etiologies.
* Subjects must have a reliable caregiver or family member who agrees to accompany the subject to all scheduled visits, provide information about the subject as required.

Exclusion Criteria:

* Subjects with any current primary psychiatric diagnosis other than dementia of the Alzheimer's type or Vascular Dementia.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2005-06; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (27):
- Canada (27):
  - Pfizer Investigational Site, Belvedere, Alberta
  - Pfizer Investigational Site, Edmonton, Alberta
  - Pfizer Investigational Site, Abbotsford, British Columbia
  - Pfizer Investigational Site, Coquitlam, British Columbia
  - Pfizer Investigational Site, Victoria, British Columbia
  - Pfizer Investigational Site, Winnipeg, Manitoba
  - Pfizer Investigational Site, Saint John, New Brunswick
  - Pfizer Investigational Site, Amherst, Nova Scotia
  - Pfizer Investigational Site, Halifax, Nova Scotia
  - Pfizer Investigational Site, Pictou, Nova Scotia
  - Pfizer Investigational Site, Burlington, Ontario
  - Pfizer Investigational Site, Corunna, Ontario
  - Pfizer Investigational Site, Fort Erie, Ontario
  - Pfizer Investigational Site, Hawkesbury, Ontario
  - Pfizer Investigational Site, North Bay, Ontario
  - Pfizer Investigational Site, Ottawa, Ontario
  - Pfizer Investigational Site, Peterborough, Ontario
  - Pfizer Investigational Site, Sarnia, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Beauport, Quebec
  - Pfizer Investigational Site, Cowansville, Quebec
  - Pfizer Investigational Site, L'Ancienne-Lorette, Quebec
  - Pfizer Investigational Site, Montreal, Quebec
  - Pfizer Investigational Site, Rimouski, Quebec
  - Pfizer Investigational Site, Saint-Jean-sur-Richelieu, Quebec
  - Pfizer Investigational Site, Saint-Léonard, Quebec
  - Pfizer Investigational Site, Regina, Saskatchewan

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2501026&StudyName=Vaspect%20Study%20-%20An%20Open-Label%20Trial%20Of%20Donepezil%20in%20Vascular%20and%20Mixed%20Dementia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted in Canada in 30 centres.
Groups:
- Donepezil: Subjects received open-label donepezil treatment with 5 mg administered per os (orally; PO)quaque die (every day; QD) for 6 weeks. Donepezil was increased to 10 mg QD (the maximum dose)at the Week-6 visit for an additional planned 18 weeks.
Period: Overall Study
Arm/Group | Donepezil
Started | 149 (148 are summarized below: 1 subject entered the study but was lost to follow up.)
Completed | 116
Not Completed | 33
Not completed — Death | 2
Not completed — Adverse Event | 19
Not completed — Withdrawal by Subject | 6
Not completed — Protocol Violation | 3
Not completed — Arrived early for last visit in error | 1
Not completed — Subject felt pill not effective enough | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Donepezil
Number analyzed (Participants) | 149
Age, Customized [Number; unit: Participants]
  < 45 | 0
  45-64 | 20
  >= 65 | 129
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82
  Male | 67

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Score of Standardized Mini-Mental State Examination (sMMSE); Full Analysis Set
Description: Change from baseline in sMMSE total score. Change: mean total score at observation minus mean total score at baseline. Total score is derived by adding all subscores and ranges from 0 to 30; a higher score indicates a better cognitive state.
Time Frame: Baseline, week 12, week 24
Population: Full Analysis Set (FAS):all subjects who received at least one dose donepezil and who have baseline and at least one post-baseline assessment of efficacy and LOCF = Last Observation Carried Forward. N=137; Weeks 12, 24 n=124, 114
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Donepezil
Number analyzed (Participants) | 137
Score on a scale
  Week 12 (n=124) | 0.41 (3.10)
  Week 24 (n=114) | 0.69 (3.2)
  Week 24 LOCF (n=137) | 0.48 (3.25)
Statistical Analysis 1: Comparison: Donepezil; Week 12 Null hypothesis; change from baseline to the final visit = 0. Alternative hypothesis; change from baseline to final visit not = to 0. Sample of 260 participants was required for study to have 85% power to detect change from baseline to final visit of 0.73 in SMMSE total score, with a SD of 3.5. Fewer than 260 patients were enrolled, due to this loss in power the number of analyses specified in the protocol has been reduced and any analyses carried out will be exploratory in nature; Test type: Superiority or Other; p = 0.182, Mixed Models Analysis — Baseline value, center, and week as fixed effects; subject was included as a random effect; Mean Difference (Net) = 0.44, 95% CI [-0.21 to 1.09], Standard Error of Mean 0.33
Statistical Analysis 2: Comparison: Donepezil; Week 24 Null hypothesis; change from baseline to the final visit = 0. Alternative hypothesis; change from baseline to final visit not = to 0. Sample of 260 participants was required for study to have 85% power to detect change from baseline to final visit of 0.73 in SMMSE total score, with a SD of 3.5. Fewer than 260 patients were enrolled, due to this loss in power the number of analyses specified in the protocol has been reduced and any analyses carried out will be exploratory in nature; Test type: Superiority or Other; p = 0.067, Mixed Models Analysis; Mean Difference (Net) = 0.66, 95% CI [-0.05 to 1.36], Standard Error of Mean 0.36
Statistical Analysis 3: Comparison: Donepezil; Week 24 LOCF Null hypothesis; change from baseline to the final visit = 0. Alternative hypothesis; change from baseline to final visit not = to 0. Sample of 260 participants was required for study to have 85% power to detect change from baseline to final visit of 0.73 in SMMSE total score, with a SD of 3.5. Fewer than 260 patients were enrolled, due to this loss in power the number of analyses specified in the protocol has been reduced and any analyses carried out will be exploratory in nature; Test type: Superiority or Other; p = 0.085, Mixed Models Analysis

2. Secondary Outcome: Disability Assessment for Dementia Change From Baseline; Activities of Daily Living (ADL) Domain.
Description: The ADL domain includes 17 yes/no questions on four items (hygiene, dressing, continence, eating). Score equals number of questions answered yes multiplied by 100 divided by number of questions answered. Change: Mean ADL score at observation minus mean ADL score at baseline.
Time Frame: Baseline, week 12, week 24
Population: Full Analysis Set (FAS): all subjects who received at least one dose of donepezil and who have baseline and at least one post-baseline assessment of efficacy and LOCF = Last Observation Carried Forward.N=137; Weeks 12, 24 n= 124, 114.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Donepezil
Number analyzed (Participants) | 137
score on a scale
  week 12 (n=124) | 1.68 (13.23)
  week 24 (n=114) | -1.61 (19.68)
  week 24 LOCF (n=137) | -1.88 (18.15)
Statistical Analysis 1: Comparison: Donepezil; Test type: Superiority or Other; p = 0.218, Mixed Models Analysis; Mean Difference (Net) = 2.0, 95% CI [-1.20 to 5.19], Standard Error of Mean 1.16
Statistical Analysis 2: Comparison: Donepezil; Test type: Superiority or Other; p = 0.385, Mixed Models Analysis; Median Difference (Net) = -1.85, 95% CI [-6.03 to 2.34], Standard Error of Mean 2.12
Statistical Analysis 3: Comparison: Donepezil; Test type: Superiority or Other; p = 0.228, Mixed Models Analysis

3. Secondary Outcome: Disability Assessment for Dementia Change From Baseline; Instrumental ADL (IADL) Domain.
Description: IADL domain consists of 23 yes-no questions on 6 items (meal preparation, telephoning, going out, finance & correspondence, medications, leisure & housework. Change: Mean IADL score at observation minus mean IADL score at baseline. Total IADL score = number of questions answered yes multiplied by 100 divided by total number of questions answered
Time Frame: Baseline, 12 weeks, 24 weeks
Population: Full Analysis Set (FAS):all subjects who received at least one dose donepezil and who have baseline and at least one post-baseline assessment of efficacy and LOCF = Last Observation Carried Forward.N=137; Weeks 12, 24 n= 124,114
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Donepezil
Number analyzed (Participants) | 137
score on a scale
  week 12 (n=124) | 1.68 (18.01)
  week 24 (n=114) | 0.20 (22.37)
  week 24 LOCF (n=137) | 1.31 (22.30)
Statistical Analysis 1: Comparison: Donepezil; Test type: Superiority or Other; p = 0.404, Mixed Models Analysis; Mean Difference (Net) = 1.84, 95% CI [-2.51 to 6.18], Standard Error of Mean 2.19
Statistical Analysis 2: Comparison: Donepezil; Test type: Superiority or Other; p = 0.826, Mixed Models Analysis; Mean Difference (Net) = 0.57, 95% CI [-4.51 to 5.64], Standard Error of Mean 2.56
Statistical Analysis 3: Comparison: Donepezil; Test type: Superiority or Other; p = 0.494, Mixed Models Analysis

4. Secondary Outcome: Disability Assessment for Dementia (DAD) Change From Baseline Total Score; Full Analysis Set (FAS)
Description: DAD total score equals total number of questions answered yes multiplied by 100 divided by total number of questions answered.
Time Frame: Baseline, week 12, week 24
Population: Full Analysis Set (FAS):all subjects who received at least one dose donepezil and who have baseline and at least one post-baseline assessment of efficacy and LOCF = Last Observation Carried Forward.N=137; Weeks 12, 24 n = 124, 114
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Donepezil
Number analyzed (Participants) | 137
score on a scale
  week 12 (n=124) | 1.71 (13.18)
  week 24 (n=114) | -0.12 (18.01)
  week 24 LOCF (n=137) | 0.17 (17.01)
Statistical Analysis 1: Comparison: Donepezil; Test type: Superiority or Other; p = 0.272, Mixed Models Analysis; Mean Difference (Net) = 1.78, 95% CI [-1.42 to 4.99], Standard Error of Mean 1.61
Statistical Analysis 2: Comparison: Donepezil; Test type: Superiority or Other; p = 0.894, Mixed Models Analysis; Mean Difference (Net) = -0.27, 95% CI [-4.21 to 3.68], Standard Error of Mean 2.00
Statistical Analysis 3: Comparison: Donepezil; Test type: Superiority or Other; p = 0.906, Mixed Models Analysis

5. Secondary Outcome: Free-hand Drawing Test (CLOX 1) Change From Baseline; Full Analysis Set (FAS)
Description: The ability to draw a clock free-hand. Scored on a scale from 1 to 15; lower scores indicate higher impairment. Change: Mean CLOX 1 score at observation minus mean CLOX score at baseline.
Time Frame: Baseline, 12 weeks, 24 weeks
Population: Full Analysis Set (FAS): all subjects who received at least one dose donepezil and who have baseline and at least one post-baseline assessment of efficacy and LOCF = Last Observation Carried Forward. N=137; weeks 12, 24 n = 123, 111
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Donepezil
Number analyzed (Participants) | 137
Score on a scale
  Week 12 (n=123) | -0.03 (3.08)
  Week 24 (n=111) | 0.95 (3.13)
  Week LOCF (n=137) | 0.74 (3.13)
Statistical Analysis 1: Comparison: Donepezil; Test type: Superiority or Other; p = 0.719, Mixed Models Analysis; Mean Difference (Net) = 0.13, 95% CI [-0.56 to 0.82], Standard Error of Mean 0.35
Statistical Analysis 2: Comparison: Donepezil; Test type: Superiority or Other; p = 0.006, Mixed Models Analysis; Median Difference (Net) = 1.00, 95% CI [0.29 to 1.71], Standard Error of Mean 0.36
Statistical Analysis 3: Comparison: Donepezil; Test type: Superiority or Other; p = 0.007, Mixed Models Analysis

6. Secondary Outcome: Copied Clock Drawing Test (CLOX 2) Change From Baseline; Full Analysis Set (FAS)
Description: The ability to copy a drawing of a clock. Scored on a scale from 1 to 15; lower scores indicate higher impairment. Change: Mean CLOX 2 score at observation minus mean CLOX 2 score at baseline.
Time Frame: Baseline, 12 weeks, 24 weeks
Population: Full Analysis Set (FAS): all subjects who received at least one dose donepezil and who have baseline and at least one post-baseline assessment of efficacy and LOCF = Last Observation Carried Forward. LOCF N=131; weeks 12, 24 n = 117, 106
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Donepezil
Number analyzed (Participants) | 131
Score on scale
  week 12 (n=117) | 0.28 (3.35)
  week 24 (n=106) | 0.84 (2.92)
  week 24 LOCF (n=131) | 0.51 (3.09)
Statistical Analysis 1: Comparison: Donepezil; Test type: Superiority or Other; p = 0.368, Mixed Models Analysis; Mean Difference (Net) = 0.32, 95% CI [-0.38 to 1.01], Standard Error of Mean 0.35
Statistical Analysis 2: Comparison: Donepezil; Test type: Superiority or Other; p = 0.030, Mixed Models Analysis; Mean Difference (Net) = 0.72, 95% CI [0.07 to 1.37], Standard Error of Mean 0.33
Statistical Analysis 3: Comparison: Donepezil; Test type: Superiority or Other; p = 0.060, Mixed Models Analysis

7. Secondary Outcome: CLOX Differential Score Change From Baseline; Full Analysis Set (FAS)
Description: CLOX differential score equals the difference between the score for CLOX 2 and the score for CLOX 1, values range from 15 to 0, with 0 indicating perfect executive function, and a worsening with the increasing score.
Time Frame: Baseline, 12 weeks, 24 weeks
Population: Full Analysis Set (FAS): all subjects who received at least one dose donepezil and who have baseline and at least one post-baseline assessment of efficacy and LOCF = Last Observation Carried Forward.LOCF N=131; weeks 12, 24 n = 117, 106
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Donepezil
Number analyzed (Participants) | 131
Score on a scale
  week 12 (n=117) | 0.26 (3.50)
  week 24 (n=106) | -0.35 (3.31)
  week 24 LOCF (n=131) | -0.44 (3.36)
Statistical Analysis 1: Comparison: Donepezil; Test type: Superiority or Other; p = 0.516, Mixed Models Analysis; Mean Difference (Net) = 0.21, 95% CI [-0.44 to 0.86], Standard Error of Mean 0.33
Statistical Analysis 2: Comparison: Donepezil; Test type: Superiority or Other; p = 0.297, Mixed Models Analysis; Mean Difference (Net) = -0.34, 95% CI [-0.97 to 0.30], Standard Error of Mean 0.32
Statistical Analysis 3: Comparison: Donepezil; Test type: Superiority or Other; p = 0.133, Mixed Models Analysis

8. Secondary Outcome: Phonectic Fluency Total Score From Baseline; Full Analysis Set (FAS)
Description: The number of words a particpant can generate in 1 minute.
Time Frame: Baseline, 12 weeks, week 24
Population: Full Analysis Set (FAS): all subjects who received at least one dose donepezil and who have baseline and at least one post-baseline assessment of efficacy and LOCF = Last Observation Carried Forward. LOCF n=136; weeks 12, 24 n = 123, 113
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Donepezil
Number analyzed (Participants) | 136
score on scale
  week 12 (n=123) | 0.84 (2.85)
  week 24 (n=113) | 0.92 (3.38)
  week 24 LOCF (n=136) | 0.83 (3.29)
Statistical Analysis 1: Comparison: Donepezil; Test type: Superiority or Other; p = 0.020, Mixed Models Analysis; Median Difference (Net) = 0.79, 95% CI [0.13 to 1.45], Standard Error of Mean 0.33
Statistical Analysis 2: Comparison: Donepezil; Test type: Superiority or Other; p = 0.018, Mixed Models Analysis; Median Difference (Net) = 0.87, 95% CI [0.16 to 1.59], Standard Error of Mean 0.36
Statistical Analysis 3: Comparison: Donepezil; Test type: Superiority or Other; p = 0.004, Mixed Models Analysis

9. Secondary Outcome: Neuropsychiatric Inventory Questionnaire (NPI-Q) Score Change From Baseline; Full Analysis Set (FAS)
Description: NPI-Q measures severity of behavioural manifestations of dementia & the level of distress each symptom gives the main caregiver, 1 (mild), 3 (severe), 0 if symptom absent, NPI-Q also measures the caregiver distress associated with each symptom,0(no distress)to 5(very severe), total score equals sum of individual item scores & ranges from 0 to 36
Time Frame: Baseline, 12 weeks, 24 weeks
Population: Full Analysis Set (FAS): all subjects who received at least one dose donepezil and who have baseline and at least one post-baseline assessment of efficacy and LOCF = Last Observation Carried Forward. LOCF n=137; weeks 12, 24 n = 124, 114
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Donepezil
Number analyzed (Participants) | 137
Score on scale
  week 12 (n=124) | -1.06 (4.02)
  week 24 (n=114) | -1.20 (4.19)
  week 24 LOCF (n=137) | -1.19 (4.03)
Statistical Analysis 1: Comparison: Donepezil; Test type: Superiority or Other; p = 0.010, Mixed Models Analysis; Mean Difference (Net) = -1.10, 95% CI [-1.93 to -0.27], Standard Error of Mean 0.42
Statistical Analysis 2: Comparison: Donepezil; Test type: Superiority or Other; p = 0.018, Mixed Models Analysis; Mean Difference (Net) = -1.12, 95% CI [-2.05 to -0.19], Standard Error of Mean 0.47
Statistical Analysis 3: Comparison: Donepezil; Test type: Superiority or Other; p = 0.018, Mixed Models Analysis

10. Secondary Outcome: Neuropsychiatric Inventory Questionnaire Distress (NPI-Q-D) Score Change From Baseline; Full Analysis Set (FAS)
Description: The total NPI-Q-D score is equal to the sum of all indiviudal symptom distress scale scores with a range of 0 to 60
Time Frame: Baseline, week 12, week 24
Population: Full Analysis Set (FAS): all subjects who received at least one dose donepezil and who have baseline and at least one post-baseline assessment of efficacy and LOCF = Last Observation Carried Forward.LOCF n=137; weeks 12, 24 n = 124, 114
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Donepezil
Number analyzed (Participants) | 137
Score on a scale
  week 12 (n=124) | -0.95 (5.54)
  week 24 (n=114) | -1.37 (6.25)
  week 24 LOCF (n=137) | -1.08 (6.04)
Statistical Analysis 1: Comparison: Donepezil; Test type: Superiority or Other; p = 0.182, Mixed Models Analysis; Mean Difference (Net) = -0.83, 95% CI [-2.06 to 0.39], Standard Error of Mean 0.62
Statistical Analysis 2: Comparison: Donepezil; Test type: Superiority or Other; p = 0.114, Mixed Models Analysis; Mean Difference (Net) = -1.09, 95% CI [-2.44 to 0.26], Standard Error of Mean 0.68
Statistical Analysis 3: Comparison: Donepezil; Test type: Superiority or Other; p = 0.038, Mixed Models Analysis

11. Secondary Outcome: Clinical Global Impressions Severity Score (CGI-S) Clinical Global Impressions Severity Score Improvement(CGI-I)Change From Baseline, Full Analysis Set (FAS)
Description: Scale measures subject's clinical condition at baseline for severity (CGI-S) & for improvement from baseline (CGI-I). At baseline subject rated on numerical scale, 1 (not at all ill) to 7 (most extremely ill). At follow up subject rated on 7 point Likert scale from 1(very much improved) to 7(very much worse) & 4 indicates no change from baseline
Time Frame: Baseline, week 24
Population: Full Analysis Set (FAS): all subjects who received at least one dose donepezil and who have baseline and at least one post-baseline assessment of efficacy and LOCF = Last Observation Carried Forward. Subjects with Baseline = 136; week 24 n = 116; week 24 LOCF n = 136
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Donepezil
Number analyzed (Participants) | 136
Score on a scale
  Baseline (n=136) | 3.40 (0.67)
  Week 24 (n=116) | 3.32 (1.21)
  Week 24 LOCF (n=136) | 3.40 (1.19)

12. Secondary Outcome: Clinical Global Impressions Severity (CGI-S)
Description: Scale measures subject's clinical condition at baseline for severity (CGI-S) subject rated on numerical scale, 1 (not at all ill) to 7 (most extremely ill).
Time Frame: Baseline
Population: Full Analysis Set (FAS): all subjects who received at least one dose donepezil and who have baseline and at least one post-baseline assessment of efficacy and LOCF = Last Observation Carried Forward. n=number of subjects with a value
Measure: Number; unit: Participants
Arm/Group | Donepezil
Number analyzed (Participants) | 136
Participants
  Normal, not at all ill (n=136) | 2
  Borderline mentally ill (n=136) | 4
  Mildly ill (n=136) | 72
  Moderately ill (n=136) | 54
  Markedly ill (n=136) | 4
  Severely ill (n=136) | 0
  Among the most extremely ill patients (n=136) | 0

13. Secondary Outcome: Clinical Global Impressions Improvement (CGI-I)
Description: Scale measures subject's clinical condition for improvement from baseline (CGI-I)subject rated on 7 point Likert scale from 1(very much improved) to 7(very much worse) & 4 indicates no change from baseline
Time Frame: Week (wk) 24
Population: Full Analysis Set (FAS): all subjects who received at least one dose donepezil and who have baseline and at least one post-baseline assessment of efficacy and LOCF = Last Observation Carried Forward. n=number of subjects with value (Week 24 n=116; Week 24 LOCF n=136)
Measure: Number; unit: Participants
Arm/Group | Donepezil
Number analyzed (Participants) | 136
Participants
  Wk 24 Very much improved (n=116) | 3
  Wk 24 Much improved (n=116) | 27
  Wk 24 Minimally improved (n=116) | 44
  Wk 24 No change (n=116) | 21
  Wk 24 Minimally worse (n=116) | 14
  Wk 24 Much worse (n=116) | 7
  Wk 24 Very much worse (n=116) | 0
  Wk 24 LOCF Very much improved (n=136) | 4
  Wk 24 LOCF Much improved (n=136) | 27
  Wk 24 LOCF Minimally improved (n=136) | 49
  Wk 24 LOCF No change (n=136) | 30
  Wk 24 LOCF Minimally worse (n=136) | 19
  Wk 24 LOCF Much worse (n=136) | 7
  Wk 24 LOCF Very much worse (n=136) | 0

14. Secondary Outcome: Clinical Global Impressions Improvement (CGI-I) Dichotomized Response
Description: Scale measures subject's (CGI-I) rated on categorial 7 point Likert scale 1 (very much improved) to 7 (very much worse) with 4 indicating no change from baseline. A dichotomized variable was created: responder = CGI-I score of 4 or less; non-responder = CGI-I score of 5 or more
Time Frame: Baseline, week 24
Population: Full Analysis Set (FAS):all subjects who received at least one dose donepezil and who have baseline and at least one post-baseline assessment of efficacy. LOCF = Last Observation Carried Forward. Week 24 n=116; Week 24 LOCF n=136
Measure: Number; unit: Particpants
Arm/Group | Donepezil
Number analyzed (Participants) | 136
Particpants
  Week 24 Responder (n=116) | 95
  Week 24 Non-responder (n=116) | 21
  Week 24 LOCF Responder (n=136) | 110
  Week 24 LOCF Non-responder (n=136) | 26

ADVERSE EVENTS:
Arm/Group | Donepezil
Serious Adverse Events (participants affected / at risk) | 24
Other Adverse Events (participants affected / at risk) | 53
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Donepezil
Cardiac failure congestive (Cardiac disorders) | 1/148
Myocardial infarction (Cardiac disorders) | 2/148
Sick sinus syndrome (Cardiac disorders) | 1/148
Abdominal pain (Gastrointestinal disorders) | 1/148
Duodenal ulcer (Gastrointestinal disorders) | 1/148
Chest pain (General disorders) | 2/148
General physical health deterioration (General disorders) | 1/148
Labyrinthitis (Infections and infestations) | 1/148
Pneumonia (Infections and infestations) | 1/148
Pyelonephritis (Infections and infestations) | 1/148
Urosepsis (Infections and infestations) | 2/148
Accidental overdose (Injury, poisoning and procedural complications) | 1/148
Fall (Injury, poisoning and procedural complications) | 1/148
Foot fracture (Injury, poisoning and procedural complications) | 1/148
Hip fracture (Injury, poisoning and procedural complications) | 3/148
Spinal compression fracture (Injury, poisoning and procedural complications) | 1/148
Electrocardiogram QT prolonged (Investigations) | 1/148
Anorexia (Metabolism and nutrition disorders) | 1/148
Electrolyte imbalance (Metabolism and nutrition disorders) | 1/148
Failure to thrive (Metabolism and nutrition disorders) | 1/148
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/148
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/148
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/148
Cerebrovascular accident (Nervous system disorders) | 2/148
Confusional state (Psychiatric disorders) | 1/148
Hallucination (Psychiatric disorders) | 1/148
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Donepezil
Diarrhoea (Gastrointestinal disorders) | 15/148
Nausea (Gastrointestinal disorders) | 26/148
Vomiting (Gastrointestinal disorders) | 9/148
Anorexia (Metabolism and nutrition disorders) | 8/148
Dizziness (Nervous system disorders) | 11/148
Headache (Nervous system disorders) | 8/148
Insomnia (Psychiatric disorders) | 15/148

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of <60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), <12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.